CLINICAL TRIAL: NCT04377906
Title: Department of Nutrition Science, Medical Faculty, Universitas Diponegoro Semarang, Indonesia
Brief Title: The Effect High Protein-Fiber Diet With Exercise on Acylated Ghrelin and Leptin in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Etika Ratna Noer, Department of Nutrition, Medical Faculty, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ERN
Record Dates: First submitted 2020-04-21; First posted 2020-05-07 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Weight Loss; Adolescent Obesity
Keywords: high protein-fiber; acylated ghrelin; leptin
MeSH Terms: conditions — Weight Loss; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: four arm parallel group with 56 young obesity:
  1. high protein-fiber diet and exercise
  2. high protein-fiber diet
  3. exercise
  4. control
Who Masked: Participant, Investigator
Masking Description: subject with random allocation Investigator do not know the group the analysator do not know the group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Protein-Fiber and Exercise (Experimental): give 1200 Kcal with 25% protein from fish and tempeh and 30g fiber from vegetable and fruit, 3 times/day and exercise : aerobic and resistance training for 5x/week, 45 minute each sesion
  Interventions: Behavioral: Modification Lifesyle
- High Protein-Fiber (Experimental): give 1200 Kcal with 25% protein from fish and tempeh and 30g fiber from vegetable and fruit, 3 times/day
  Interventions: Behavioral: Modification Lifesyle
- Exercise (Experimental): aerobic and resistance training for 5x/week, 45 minute each sesion
  Interventions: Behavioral: Modification Lifesyle
- control (No Intervention): regular diet

INTERVENTIONS:
Behavioral: Modification Lifesyle — high protein-fiber and exercise
  Arms: Exercise; High Protein-Fiber; High Protein-Fiber and Exercise

SUMMARY:
Obesity has been reported to impair regulation of appetite and lead uncontrollably hunger and satiety response. Ghrelin is orexigenic hormone from the stomach meanwhile, leptin is anorexigenic from adipose. Interestingly, obesity is associated with acylated ghrelin and leptin resistance. Study about the impact of high protein and fiber with combined exercise (HPFE) to suppress hunger among young obese still unclear. The hypothesis was that high protein-fiber would result in decreased in acylated ghrelin and leptin in HPFE group. Thus, the investigator examined the effect of an 8 weeks HPFE on acylated ghrelin and leptin. Subjects were randomized into four groups: High Protein-Fiber (HPF; n=15). High Protein-Fiber and exercise (HPFE; n=15), Exercise (E; n=15) and control (C; n=15). The diet prescribed 1200 kcal/day, based on basic energy requirement minus 300kcal, consisted high protein (25%) and fiber (30g/day). The exercise is combination aerobic and resistance training, with target 75% heart rate maximum. Plasma acylated ghrelin and leptin were analyzed with enzyme immunoassay.

DETAILED DESCRIPTION:
1. Introduction Obesity pandemic occurred in both developed and developing countries. The prevalence of young obesity is rising among adolescents in developing countries as well, rising from 8.1% to 12.9% in 2013 for boys and from 8.4% to 13.4% in girls. The Indonesian Basic Health Research showed prevalence of young obesity in Indonesia increase from 18,8 menjadi 31% on 2007 till 2018. The prominent problem with young obesity is the accumulation of adipose cells in the abdominal which can interfere with appetite hormones. Ghrelin is the only known as orexigenic hormon which secreted from the stomach. The leptin is one of anorexigenic mainly released by the adipose tissue. The orexigenic hormone acylated ghrelin and the anorexigenic hormones leptin are an important players in regulating appetite, food intake, energy balance, and adipogenesis.

   Regarding body weight regulation, key element are the control of energy intake which is regulated at the simplest level by sensation of hunger. Body weight is controlled by a complex system, including both peripheral and central factors. Two of the hormones that appear to play a crucial role in the regulation of food intake and body weight are leptin and ghrelin. Interestingly, obesity is associated with acylated ghrelin and leptin resistance. Hyperleptinemia is blunted response in satiety. Postprandial acylated ghrelin levels in obesity abdominal subjects do not fall, so hunger still appears. In obese subjects experience leptin resistance because the leptin receptor is disrupted so that there is a failure of sending leptin signals to the hypothalamus. Many study especially about acylated ghrelin still controversial. Studi Andarini showed plasma AG concentration is higher before and after eating at all time points, regardless of food type, in obese individuals, as compared with normal weight individuals. Consistant with the Ozkan et al reveal the AG increase following obesity status.

   Different types of protein can result in different levels of satiety. Metabolites, including certain amino acids, contribute to the food intake is arginine. The ability of specific L-amino acids, including L-arginine (L-Arg), to stimulate anorectic agent (GLP-1 and PYY) release has been studied previously in vitro. The study Alamshah et al showed L-Arg reduced food intake and stimulated gut hormone release in rodents. The role fiber affect the release satiety and gastric emptying rate.

   Managing weight loss with modification lifestyle in young obesity actually requires paying special attention to high compliance and less hunger more satiety. The study aimed to examine the effect of giving a high protein diet rich arginine and fiber diet with exercise among adolescent obesity.
2. Methods and Matherials 2.1 Participants The program was conducted from Juli to Oktober 2018. Subject were recruited through nutrition screening and campaign mass media. For sample size, the investigator calculated previous studies regarding AG with following setting: power was set at 80%, p value at 0.5 and standardized difference was 21.2, resulting in a sampel size of 12 subjects, including 20% for drop out. Inclusion criteria are body mass index > 25 kg/m2, waist circumference >80 cm for female and >90 cm for male. The investigator exclude who were taking dietary supplements or medication, smokers, have pregnancy, lose body weight > 10% before treatment and have chronic disease history. The participants consisted of 60 adolescents obesity who were selected from outpatient of Universitas Diponegoro, Semarang, Indonesia. Subjects were randomized into four groups : High Protein-Fiber (HPF; n=15). High Protein-Fiber and exercise (HPFE; n=15), Exercise (E; n=15) and control (C; n=15). All participants has signed informed consent and the study was approved by Kariadi Hospital-Diponegoro University with provision Declaration of Helsinki (Number 427/EC/FK-UNDIP/VII/2018)

2.1 Study design and randomization. The study design was randomized clinical trial (four-arm). The random assignment was generated by a computerized program. The duration of intervention is 8 weeks. It was not possible to blind the dietitians who advised on dietary prescribe.

3.1 Diet protocol The subject were randomly into four of different intervention. The HPFE prescribed balanced diet (55%carbohydrate, 25% protein, and 20% fat). Based on the Academy Dietetics of Association recommends using the Miflin-St Jeor equation for estimating RMR in obese individuals. Subject have body weight means 75 kg, so the total energy was calculated 1500 kcal,then minus 300kcal. The distribution energy of breakfast (30%), lunch (40%) and dinner (30%) and extra 500ml plan water before meal. The investigator choose the protein sources rich arginine like all type fish, tempeh, nuts/peas. The investigator serve the diet menu everyday in our laboratory. The diet was prescribed with the use of standardazied household measure to quatify the food portion in each meal. The subjects were monitored the diet everyday with logbook. The control group give nutrition education once a week in nutrition laboratory. The nutritional data was calculated by software (Nutrisurvey).

4.1 Exercise protocol

One session of training program included the following program component :

1) 5 min warm-up; 2) 25 min aerobic training; 3) 10 min resistance training, 4) 5 min cool-down. The resistance training was performed without weight training machine (chalestenic). The movement includes plank, mountain climber, pilates leg pulls, right side plank, left side plank, flutter kick, toe touch crunches, crunch, knee tuck crunches and russian twist. The muscle strength level by 40 repetition maximum (RM). Rest between the sets of the resistance training was set 20reps. The aerobic training was performed koreographic for at least 25 min and the intensity was 75% heart rate maximum. The frequency of training was five times a week (on alternate day) under professional trainer. Heart rate during training was monitored using HR monitor (H10, POLLAR, Kemple, Finland)

5.1 Body composition Body weight, and percent body fat mass, were analyzed by a bioelectric impedance analyzer (TANITA DC-360) with light clothes and no shoes. Height was measured by stadiometer (SECA 207). BMI was calculated as body weight in kilograms divided by height in meters squared (kg/m2). Waist Circumference (WC) was measured with a inelastic measuring tape around the mid-section between the margin of the last rib and the iliac crest.

6.1 Hormone Analysis Venous blood samples were obtain after 10h fasting. Blood samples for insulin and leptin were stored in plain tubes, and acylated ghrelin were stored in tubes with EDTA. For active ghrelin, immediately after collection, 40 mL p-hydroxymercuribenzoic acid was added to each blood sample. The samples were centrifuged at 3500X at 4C for 10 min. For acyl ghrelin, after centrifugation, the plasma was pipetted in 1.5-mL microtubes, and 100 mL hydrochloric acid (1N) was added for each 1 mL plasma. For all blood sample, the respective supernatant fluids were pipetted and frozen at 80°C for a later analysis by an enzyme-linked immunoassay (Elabscience E-EL-H2002 for AG, E-EL-H0113 for leptin). Blood samples for trigliserida and HDL were stored in tubes with non EDTA, and analyzed with clinical chemistry automatic analyzer (Indiko thermoscientific).

7.1 Statistical Analysis Data were analyzed IBM SPSS. Variable not normally distributed were nonparametric test. Wann whitney U test was used to test for difference all parameter at baseline. We compared change in variable (baseline-week8) in each sub group using pair t=test or wilcoxon signed rank test to determine the impact of differential change. To test for change in parameters between four group used kruskal wallis.

ELIGIBILITY:
Inclusion Criteria:

* body mass index > 25 kg/m2,
* waist circumference >80 cm for female and >90 cm for male

Exclusion Criteria:

* taking dietary supplements or medication
* smokers
* have pregnancy
* lose body weight > 10% before treatment
* have chronic disease history

Ages: 19 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female and male is equal
Enrollment: 56 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
change acylated ghrelin | 8 weeks
  Change from Baseline acyl ghrelin at 8 weeks taken in the lab from venous blood specimen after10h fasting using ELISA method
change leptin | 8 weeks
  Change from Baseline leptin at 8 weeks taken in the lab from venous blood specimen after10h fasting using ELISA method
change body weight | 8 weeks
  change from baseline body weight at 8 weeks measured using bioelectrical impedance analysis (BIA) with light clothes and no shoes

SECONDARY OUTCOMES:
change triglyceride | 8 weeks
  change from baseline triglyceride at 8 weeks taken in the lab from venous blood specimen after10h fasting
change high density lipoprotein | 8 weeks
  change from baseline high density lipoprotein at 8 weeks taken in the lab from venous blood specimen after10h fasting

CONTACTS AND LOCATIONS:
Overall Officials: Etika Noer, Principal Investigator — Diponegoro University
Locations (1):
- Etika Ratna Noer, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
the result of this study is available to cite everyone
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: etikaratna@fk.undip.ac.id
URL: http://dept-gizi@fk.undip.ac.id